CLINICAL TRIAL: NCT01237782
Title: Efficacy of a Propolis Solution for Cleaning Complete Dentures: a Randomized Crossover Trial
Brief Title: Efficacy of a Propolis-based Denture Cleanser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raphael Freitas de Souza (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Raphael Freitas de Souza, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FORP-PT-002; 2009.1.1081.58.6 (Other: Institutional Review Board (FORP-USP)); 2009/53788-9 (Other Grant/Funding Number: FAPESP (São Paulo Research Foundation))
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Dental Plaque; Denture Stomatitis; Oral Candidiasis; Oral Hygiene
Keywords: Candida; Complete Denture; Dental Plaque Index; Denture Bases; Denture Cleansers; Edentulous Mouth; Mutans Streptococci; Oral Health; Propolis; Streptococcus mutans
MeSH Terms: conditions — Dental Plaque; Stomatitis, Denture; Candidiasis, Oral; Torulopsis; Mouth, Edentulous | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propolis solution (Experimental): A proprietary denture cleanser with propolis as the active agent.
  Interventions: Drug: Denture soaking solution
- Saline solultion (Placebo Comparator): Physiologic saline solution.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Denture soaking solution — Immersion of complete dentures in 200ml of a denture soaking solution for 20 minutes. Propolis solution: Spa Dent (Nissin Dental Products Inc., Kyoto, Japan).
  Other Names: Chemical methods for cleaning dentures; Chemical dentures cleaners; Crude drugs; Propolis denture cleaner; Propolis solution
  Arms: Propolis solution
Drug: Saline solution — Immersion of complete dentures in 200ml of a placebo denture soaking solution for 20 minutes.
  Arms: Saline solultion

SUMMARY:
The purpose of this study is to assess if a propolis solution is able to remove plaque and kill microbes from complete dentures. The investigators will compare the results of the propolis-based denture cleanser with those obtained with an inactive solution.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Patients requesting new complete dentures
* Regular wearing of the same maxillary and mandibular complete dentures for at least one year
* Both denture bases and artificial teeth should be composed by acrylic resin

Exclusion Criteria:

* Unsatisfactory complete dentures in use (i.e. with poor fitting, relining or fractures)
* Pathologic changes in the oral cavity

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Denture plaque coverage area (%) | At the same day of the intervention, up to 1 hour following denture soaking
  Relation between stained area and total surface area on the internal surface of maxillary complete dentures.

SECONDARY OUTCOMES:
mutans streptococci counts (CFU) | At the same day of the intervention, up to 1 hour following denture soaking
  Microbial counts on maxilary denture base, as assessed by a conventional microbiological method.
Candida spp. counts (CFU) | At the same day of the intervention, up to 1 hour following denture soaking
  Microbial counts on maxilary denture base, as assessed by a conventional microbiological method.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael F de Souza, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Ribeirão Preto Dental School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Institutional page of the Ribeirão Preto Dental School (research site) — http://www.forp.usp.br
- See also: Principal Investigator´s CV — http://sistemas3.usp.br/tycho/CurriculoLattesMostrar?codpub=F7A61880194F